CLINICAL TRIAL: NCT04044846
Title: Promoting Movement in Older Adults in the Community
Acronym: (ProMO)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID-19 pandemic caused several challenges with recruitment in the home care sector. It was not possible to proceed with the study as originally intended in this clinical trial record.
Sponsor: Regional Geriatric Program of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 239-2019
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Frailty; Mobility Limitation
MeSH Terms: conditions — Frailty; Mobility Limitation

STUDY DESIGN:
Intervention Model Description: The pilot evaluation will have a quasi-experimental pre-test/post-test design and investigators will collect self- reported data from frail older adults on the perceived benefit of exercise using the Vitality Plus Scale (VPS) (Myers et al., 1999).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The recipients of the home-based physical activity program (Experimental): Frail OAs will be asked to fill out the Vitality Plus Scale at the beginning of the implementation phase (baseline) by a research assistant over the telephone. At the end of the 6-month implementation phase, the research assistant will administer the survey again (post-intervention).
  Interventions: Behavioral: Physical activity program for homebound older adults faciliated by Personal Support Workers

INTERVENTIONS:
Behavioral: Physical activity program for homebound older adults faciliated by Personal Support Workers — The intervention is an evidence- informed, theory-driven mobility intervention for community-dwelling OAs who are moderately and severely frail according to the clinical frailty scale (Rockwood et al., 2005). The intervention, entitled Promoting Movement in OAs (ProMO), will be implementable with frail OAs in partnership with any care provider in the home. Investigators will focus the study on the two main providers of care- personal support workers (PSWs) and family caregivers. OAs, PSWs, and caregivers will co-create ProMO with us. ProMO will be distinct from existing home-based exercise programs (Johnson et al., 2003) (Giangregorio et al., 2018) because it will optimize natural opportunities for mobilization during care (e.g., bathing and dressing) and will be embedded in facilitated activities of daily living.
  Other Names: ProMO

SUMMARY:
It is well known that exercise is great medicine, however, for frail older adults who are often homebound and require assistance with personal care, there are gaps in both prescribing this "medicine" and in filling the prescription. The investigators will uncover and address the barriers that prevent frail older adults from increasing their level of physical activity. With input from frail older adults, caregivers, and healthcare providers, the investigators will create a free, easy to use, home-based program that incorporates physical activity such as gentle stretches and range of motion exercises when personal care is being provided. This innovation will add great value to the type of care that is being provided to homebound frail older adults. Incorporating physical activity as part of the care provided offers a unique opportunity for homebound frail older adults to move more, and improve their well-being.

DETAILED DESCRIPTION:
Mobilization in frail older adults (OAs) can improve cardiovascular outcomes, musculoskeletal function, and functional independence (Bray, Smart, Jakobi, & Jones, 2016) (Roland, Theou, Jakobi, & Frailty, 2014) (Theou et al., 2011). Detriments of immobility include an increased risk of functional disability, falls, and premature mortality (Hubbard, Parsons, Neilson, & Carey, 2009). There are numerous mobility interventions targeted to community-dwelling frail OAs (Sherrington et al., 2019); however, they either have a narrow focus on falls prevention (Fairhall, Sherrington, & Cameron, 2013) (Sherrington et al., 2019) or they target mildly frail OAs (Johnson, Myers, Scholey, Cyarto, & Ecclestone, 2003) (Giangregorio et al., 2018) (Binder et al., 2002). A review of home-based mobility interventions concluded that high-risk OAs who have been recently discharged from hospital may require an intervention that is tailored specifically for them (Hill, Hunter, Batchelor, Cavalheri, & Burton, 2015) (Sherrington et al., 2019). The intervention will focus on active range of motion exercises in frail OAs who are homebound or recovering from a health crisis and unable to participate in more rigorous exercise regimens. Gentle stretches and range of motion activities can have immediate benefits to frail OAs. (O'Brien Cousins & Horne, 1999).

The first objective is to create an evidence- informed, theory-driven mobility intervention for community-dwelling OAs who are moderately and severely frail according to the clinical frailty scale (Rockwood et al., 2005). The intervention, entitled Promoting Movement in OAs (ProMO), will be implementable with frail OAs in partnership with any care provider in the home such as personal support workers (PSWs) and families. The investigators will focus the study on the two main providers of care- PSWs. OAs, PSWs, and caregivers will co-create ProMO with us. ProMO will be distinct from existing home-based exercise programs (Johnson et al., 2003) (Giangregorio et al., 2018) because it will optimize natural opportunities for mobilization during care (e.g., bathing and dressing) and will be embedded in facilitated activities of daily living. The second objective is to pilot and evaluate ProMO in the Greater Toronto Area (GTA). The primary output will be a free, user-friendly, and sustainable mobility intervention. A secondary output will be new knowledge about the process and outcome of a tailored, home-based mobility intervention.

ELIGIBILITY:
Inclusion Criteria:

* Older adults living with frailty who are homebound and using home care services.

Exclusion Criteria:

* Older adults who are not living with frailty and not homebound.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Perceived benefit of exercise | 6 months
  The 10-item Vitality Plus Scale (VPS) was developed to measure the health-related benefits of mobilization specifically in OAs. It is a self-administered, 10-item scale, which assesses multiple domains, including sleep, energy, pain and mood. Participants will be asked to provide a rating from 1 to 5 for each of the 10 items. A total score will be calculated for each individual and a total score can range from 1 to 50. A 10% increase in VPS score was considered clinically significant for an individual. The investigators hypothesize that the intervention will result in an increase in post VPS scores. The VPS has been shown to be reliable and valid, sensitive to change and easy for OAs to use. It has been used to measure the effects of mobilization in randomized controlled trials (Li et al., 2013) (Burton, Lewin, Clemson & Boldy, 2013) (Chin A Paw, van Poppel, Twisk & van Mechelen, 2004) (Stiggelbout, 2004).

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Geriatric Program of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared with other researchers.